CLINICAL TRIAL: NCT03748095
Title: Population Pharmacokinetic Modeling to Optimize the Dosage of the Piperacillin / Tazobactam Combination in Patients With Sepsis in Intensive Care
Acronym: OPT-TAZ
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02681-54; 2017/384/HP (Registry Identifier: CHU Rouen)
Record Dates: First submitted 2018-11-16; First posted 2018-11-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Resuscitation Patients With Sepsis
MeSH Terms: interventions — Piperacillin; Tazobactam

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: pipéracilline/tazobactam — There is not intervention description

SUMMARY:
Population pharmacokinetic modeling mathematically describes the pharmacokinetics of a drug and the variables likely to influence it in a "typical" patient population. We propose to model a Bayesian estimator, taking into account the individual factors that influence exposure to the piperacillin / tazobactam combination in a target population of sepsis, to allow for early assessment of serum Piperacillin / Tazobactam concentration profiles. optimization of dosing regimens. Indeed, pharmacokinetic tools of this type are already regularly successfully applied for other classes of antibiotics or immunosuppressants whose therapeutic index is narrow. They reduce the toxic risk and optimize the effectiveness of these treatments.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (age ≥18 years) male or female.
* Patient hospitalized in intensive care for sepsis, involving (i) a suspected or proven infection; (ii) a systemic inflammatory response; (iii) dysfunction of at least one organ, according to the international consensus "sepsis-3".
* Patient with an arterial catheter that can be used for blood sampling by the time the first dose of piperacillin / tazobactam is administered.
* Patient for whom treatment with piperacillin / tazobactam, alone or in combination with another antibiotic, is prescribed according to the following modalities (drug SPC): scheduled antibiotic treatment for at least 48 hours in IV infusion of 4 g of piperacillin and 0.5 g tazobactam over 3 hours, every 6 hours or every 8 hours.
* Patient affiliated to a social security scheme.
* Patient informed and given his non-opposition. If the patient is unable to do so (emergency situations) the non-opposition will be obtained from the patient's representative.

Exclusion Criteria:

* Treatment with piperacillin and / or tazobactam within 7 days prior to evaluation.
* Patient with a history of allergy to penicillins or β-lactams.
* Kidney function of Kdigo score = 3 (3 times baseline plasma creatinine or plasma creatinine ≥ 354μmol / L or extra-renal clearance, or diuresis <0.3ml / kg / h for ≥ 24h or anuria for ≥ 12h) to not include patients at very high risk of extra-renal clearance within 48 hours.
* Hypersensitivity to the active substances, to any other antibacterial agent of the penicillin class or to any of the excipients.
* History of severe allergic reaction to any other β-lactam.
* Patient being treated with extrarenal treatment.
* Patient being treated with extracorporeal circulation (ECMO).
* Hepatic insufficiency patient with Child C. cirrhosis.
* Patient who refused to participate or refused participation by the representative.
* Person deprived of liberty by an administrative or judicial decision.
* Person under tutorship or curatorship.
* Pregnant or nursing woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalized in intensive care for sepsis, involving (i) a suspected or proven infection; (ii) a systemic inflammatory response; (iii) dysfunction of at least one organ, according to the international consensus "sepsis-3"
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-03-12 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
The objective is to develop a Bayesian estimator of the area under the blood concentration curves of the piperacillin / tazobactam combination in resuscitation patients with sepsis. | 24hours
  The primary endpoint of this study is the ability of the pharmacokinetic model developed to predict the AUC of the piperacillin / tazobactam combination at 24 hours after initiation of antibiotic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rouen, Rouen, France

IPD SHARING:
Plan to Share IPD: No